CLINICAL TRIAL: NCT01871103
Title: The Dorsal Homodigital Island Flap Based on the Dorsal Branch of the Digital Artery: A Review of 171 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HBTS1306017
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2007-01

CONDITIONS: Soft Tissue Defect; Sensory Reconstruction of Digits; Multiple Digital Defects
Keywords: Soft tissue defect; dorsal branch of the digital artery; dorsal branch of the digital nerve; dorsal homodigital island flap

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical flap (Other): The dorsal homodigital island flap is a perforator type flap based on the DB, which uses the dorsal skin of the injured finger to provide soft tissue coverage for a volar defect.
  Interventions: Procedure: The dorsal homodigital island flap

INTERVENTIONS:
Procedure: The dorsal homodigital island flap — The dorsal homodigital island flap is used for tissue reconstruction in different regions of the finger.

SUMMARY:
Soft tissue reconstruction in the finger continues to evolve. The dorsum of the finger is a reliable flap donor site in reconstructive hand surgery because of its similar quality to the original. The dorsal homodigital island flap can be used as a reliable alternative for reconstructing small to moderate defects of the fingers. In this retrospective study, the investigators would evaluate the efficacy of the technique for tissue reconstruction in different regions of the finger, with an emphasis on sensibility, pain and donor site morbidity.

DETAILED DESCRIPTION:
At final follow-up, sensory restoration of the flap is measured using the static 2-point discrimination test and Semmes-Weinstein monofilament test. We evaluate pain sensations of the reconstructed fingers and donor sites with a visual analog scale. The system consist of a 10 cm line that is grouped into mild (0-3 cm), moderate (4-6 cm) and severe (7-10 cm). Active motion of the joints is measured using a goniometer. The motion arcs of the reconstructed fingers are compared with the opposite side.

ELIGIBILITY:
Inclusion Criteria:

* the soft tissue defect in one finger or in multiple fingers
* a defect > 1.5 cm and < 3 cm in length
* necessity to preserve finger length
* a patient between 15 and 60 years of age

Exclusion Criteria:

* injuries to the dorsum of the finger or to the course of the vascular pedicle that precluded its use as the donor
* a defect≤1.5 cm or ≥3 cm in length
* a soft tissue defect of the thumb

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Static 2-point discrimination test | 18 months to 24 months
  The test point is at the center of the flap. Each area was tested 3 times with a Discriminator (Ali Med, Dedham, MA). We stop at 4mm as a limit of 2PD and considered this normal.

SECONDARY OUTCOMES:
Cold intolerance | 18 months to 24 months
  We access the cold intolerance of the injured and donor fingers using the self-administered Cold Intolerance Severity Score questionnaire10 that is rated into mild, moderate, severe, and extreme (0-25, 26-50, 51-75 and 76-100).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Tang P, Zhang X. Sensory reconstruction of a finger pulp defect using a dorsal homodigital island flap. Plast Reconstr Surg. 2012 Nov;130(5):1077-1086. doi: 10.1097/PRS.0b013e318267ef99. PMID 22777035
- [Derived] Chen C, Tang P, Zhang X. The dorsal homodigital island flap based on the dorsal branch of the digital artery: a review of 166 cases. Plast Reconstr Surg. 2014 Apr;133(4):519e-529e. doi: 10.1097/PRS.0000000000000016. PMID 24675204